CLINICAL TRIAL: NCT07242365
Title: A Phase II Study Integrating Soylent™ Meal Replacement to Reduce Gastrostomy Tube Rates in Patients With Head &Amp; Neck Cancer Undergoing Chemoradiotherapy
Brief Title: Soylent in Reducing Gastrostomy Tube Rates in Patients With Locally Advanced Head and Neck Cancer Undergoing Chemoradiotherapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-000033; NCI-2017-01225 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17-000033 (Other: UCLA / Jonsson Comprehensive Cancer Center); P30CA016042 (NIH)
Record Dates: First submitted 2023-10-13; First posted 2025-11-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Head and Neck Carcinoma
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (Soylent) (Experimental): Patients receive Soylent PO for up to 3 months.
  Interventions: Dietary Supplement: Soylent Graham Dietary Supplement; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Dietary Supplement: Soylent Graham Dietary Supplement — Given Soylent PO
  Other Names: Dietary Supplement; Dietary Supplements; Nutritional Supplement; Supplement; supplemental nutrition; Supplements
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies Soylent in reducing gastrostomy tube rates in patients with head and neck cancer that has spread to nearby tissues or lymph nodes (locally advanced) who are undergoing chemoradiotherapy. Soylent is a liquid meal replacement product that may reduce the risk of malnutrition and gastrostomy placement during or following treatment for head and neck cancer with chemoradiation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the compliance rate of oral nutritional replacement with Soylent.

II. To determine the overall therapeutic gastrostomy (G)-tube placement rate (G-tube placement from the 1st day of chemoradiation up to 4 weeks following treatment).

SECONDARY OBJECTIVES:

I. To determine weight loss and body mass index (BMI) changes during and following treatment.

II. To determine the change in nutritional and metabolic biomarkers during treatment.

III. To determine physician-reported acute and late toxicities during and following treatment.

IV. To determine patient-reported quality of life during and following treatment.

V. To determine clinical outcomes from treatment.

OUTLINE:

Patients receive Soylent orally (PO) for up to 3 months.

After completion of study, patients are followed up at 1, 3, 6, 12, 16, 18 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented locally advanced head and neck malignancies for which concurrent chemoradiation has been recommended for definitive or adjuvant treatment
* No history of prior radiotherapy to the head and neck; however, if previous treatment was superficial skin radiotherapy without regional lymph node treatment this will be allowed
* Karnofsky performance status (KPS) >= 70
* Body mass index >= 18 kg/m^2
* No evidence of metastatic disease (M1 disease)
* No G-tube placement prior to initiation of chemoradiation
* Eligible to undergo concurrent chemotherapy as determined by treating medical oncologist
* If a woman is of childbearing potential, a negative serum pregnancy test must be documented prior to proceeding with chemoradiation; women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) for at least 4 weeks after study treatment
* Ability to understand and willingness to sign a written informed consent
* Able to tolerate the taste of one of the flavors of the oral nutritional supplement Soylent
* Able and willing to participate in the Swallow Preservation Program at the Speech Pathology Clinic
* No evidence of clinically significant swallowing dysfunction by history or physical exam at time of radiation oncology consultation

Exclusion Criteria:

* Patients who have previously received therapeutic radiation therapy to the head and neck except for superficial skin radiotherapy is allowed
* Patients who had G-tube placement due to concern for aspiration or due to severe malnutrition in advance of chemoradiation
* Patients underweight in advance of chemoradiation (BMI < 18 kg/m^2)
* Patients who refuse to use Soylent oral nutritional supplementation due to its taste or other patient preference reasons
* Patients with allergies to any of the ingredients contained in the nutritional supplement
* Pregnant women, or women of childbearing potential who are sexually active and not willing/able to use medically acceptable forms of contraception for the entire study period and for up to 4 weeks after the study treatment
* Refusal to sign the informed consent
* Refusal to participate in the Swallow Preservation Program prior to start of Soylent if applicable
* Evidence of clinically significant swallowing dysfunction by history or physical exam at time of radiation oncology consultation
* Distant metastatic disease (M1 disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-06-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Compliance with Soylent nutritional supplementation | Up to 24 months
  The compliance rate and the corresponding 95% exact confidence interval will be calculated.
Therapeutic gastrostomy (G)-tube placement rate | Up to 24 months
  The G-tube placement rate will be analyzed using one-sample exact binomial test. The 95% exact confidence interval will be provided.

SECONDARY OUTCOMES:
Weight change | Up to 24 months
  Will be collected at each visit and summary descriptive statistics will be calculated at each time points. Repeated measure analysis of variation will be used to explore if there are any change in these parameters over time.
Body mass index | Up to 24 months
  Will be collected at each visit and summary descriptive statistics will be calculated at each time points. Repeated measure analysis of variation will be used to explore if there are any change in these parameters over time.
Treatment breaks | Up to 24 months
  Will be recorded in days per study patient and summarized.
Timing and duration of G-tube placement | Up to 24 months
  G-tube placement timing will be recorded for patients receiving G-tubes, and the duration of G-tube dependence will be recorded in days per study patient and summarized.
Serum human papilloma virus deoxyribonucleic acid | Up to 24 months
  Will be summarized by descriptive statistics by visit time points, and these statistics will be plotted graphically.
Pre-albumin | Up to 24 months
  Will be summarized by descriptive statistics by visit time points, and these statistics will be plotted graphically.
Albumin | Up to 24 months
  Will be summarized by descriptive statistics by visit time points, and these statistics will be plotted graphically.
C-reactive protein | Up to 24 months
  Will be summarized by descriptive statistics by visit time points, and these statistics will be plotted graphically.
Interleukin-6 | Up to 24 months
  Will be summarized by descriptive statistics by visit time points, and these statistics will be plotted graphically.
Tumor necrosis factor | Up to 24 months
  Will be summarized by descriptive statistics by visit time points, and these statistics will be plotted graphically.
Vitamin A | Up to 24 months
  Will be summarized by descriptive statistics by visit time points, and these statistics will be plotted graphically.
Vitamin C | Up to 24 months
  Will be summarized by descriptive statistics by visit time points, and these statistics will be plotted graphically.
Vitamin D | Up to 24 months
  Will be summarized by descriptive statistics by visit time points, and these statistics will be plotted graphically.
Tryptophan | Up to 24 months
  Will be summarized by descriptive statistics by visit time points, and these statistics will be plotted graphically.
Kynurenine | Up to 24 months
  Will be summarized by descriptive statistics by visit time points, and these statistics will be plotted graphically.
Leptin | Up to 24 months
  Will be summarized by descriptive statistics by visit time points, and these statistics will be plotted graphically.
Adiponectin | Up to 24 months
  Will be summarized by descriptive statistics by visit time points, and these statistics will be plotted graphically.
Complete metabolic panel | Up to 24 months
  Will be summarized by descriptive statistics by visit time points, and these statistics will be plotted graphically.
Complete blood count | Up to 24 months
  Will be summarized by descriptive statistics by visit time points, and these statistics will be plotted graphically.
Radiosensitivity biomarker panel | Up to 24 months
  Will be summarized by descriptive statistics by visit time points, and these statistics will be plotted graphically.
Incidence of physician-reported acute and late toxicities | Up to 24 months
  Toxicity will be graded using the Common Toxicity Criteria for Adverse Events version 4.0. Adverse events and serious adverse events will be reported using a Common Terminology Criteria for Adverse Events version 4.0 terminology and severity.
University of Washington and Functional Assessment of Cancer Therapy questionnaire assessment of Patient-reported quality of life | Up to 24 months
  Will be summarized by descriptive statistics by visit time points.
Local/loco-regional control | Up to 24 months
  Will be estimated using the Kaplan-Meier method.
Distant metastasis-free survival | Up to 24 months
  Will be estimated using the Kaplan-Meier method.
Overall survival | Up to 24 months
  Will be observed.

CONTACTS AND LOCATIONS:
Overall Officials: John Hegde, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States